CLINICAL TRIAL: NCT06699485
Title: Short-term Effects of Carbohydrate-restricted Diet on Glycemic and Metabolic Control Among Children and Adolescent With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadeer Soliman Kamaleldin, Resident of pediatric department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-15-10-1MS
Record Dates: First submitted 2024-11-16; First posted 2024-11-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Children and adolescents aged 10 - 18 years, diagnosed with T1DM for at least 1 year
  Interventions: Dietary Supplement: Low carb diet

INTERVENTIONS:
Dietary Supplement: Low carb diet — Low-carbohydrate diet contains (<26% carbohydrates) or less than 130 g/d

SUMMARY:
The current management of type 1 diabetes mellitus (T1DM) involves the use intensive insulin therapy, frequent blood glucose monitoring and carbohydrate counting.

There is a need to strengthen some of the T1DM management aspects as dietary intervention in order to achieve better glycemic and metabolic control.

The international society for pediatric and adolescent diabetes (ISPAD) recommend that children and adolescents with T1DM have about 50% of their total daily caloric requirement from carbohydrates. However, an alternative approach is emerging in recent years. The use of low-carbohydrate diet is suggested to reduce postprandial hyperglycemia and glycemic variability and lower the required insulin.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10 - 18 years, diagnosed with T1DM for at least 1 year attending the Pediatric diabetes clinic at Sohag University Hospital and using the MDI regimen and carbohydrate counting methods are eligible for the study.

Exclusion Criteria:

* Children and adolescents with associated diseases such as autoimmune hypothyroidism or celiac disease and those with diabetes-related complications such as diabetic neuropathy, retinopathy or nephropathy will be excluded.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
The blood glucose level | 6 months
  The blood glucose levels will be measured for the study participants by finger-stick glucometer

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag universty hospital, Sohag, Egypt

REFERENCES:
- [Background] Bravata DM, Sanders L, Huang J, Krumholz HM, Olkin I, Gardner CD, Bravata DM. Efficacy and safety of low-carbohydrate diets: a systematic review. JAMA. 2003 Apr 9;289(14):1837-50. doi: 10.1001/jama.289.14.1837. PMID 12684364
- [Background] Mitsui Y, Kuroda A, Ishizu M, Mori H, Kurahashi K, Kondo T, Yoshida S, Akehi Y, Aihara KI, Endo I, Abe M, Matsuhisa M. Basal insulin requirement in patients with type 1 diabetes depends on the age and body mass index. J Diabetes Investig. 2022 Feb;13(2):292-298. doi: 10.1111/jdi.13547. Epub 2021 May 3. PMID 33740836
- [Background] Kuroda A, Yasuda T, Takahara M, Sakamoto F, Kasami R, Miyashita K, Yoshida S, Kondo E, Aihara K, Endo I, Matsuoka TA, Kaneto H, Matsumoto T, Shimomura I, Matsuhisa M. Carbohydrate-to-insulin ratio is estimated from 300-400 divided by total daily insulin dose in type 1 diabetes patients who use the insulin pump. Diabetes Technol Ther. 2012 Nov;14(11):1077-80. doi: 10.1089/dia.2012.0109. PMID 23101953
- [Background] Abraham MB, Jones TW, Naranjo D, Karges B, Oduwole A, Tauschmann M, Maahs DM. ISPAD Clinical Practice Consensus Guidelines 2018: Assessment and management of hypoglycemia in children and adolescents with diabetes. Pediatr Diabetes. 2018 Oct;19 Suppl 27:178-192. doi: 10.1111/pedi.12698. No abstract available. PMID 29869358